CLINICAL TRIAL: NCT06129955
Title: A Phase II Clinical Study on the Efficacy and Safety of Pucotenlimab Combined With Lenvatinib as a Neodjuvant Therapy for Non Clear Cell Renal Cell Carcinoma With Indications for Partial Nephrectomy But High Surgical Risk: A Single Arm Approach
Brief Title: Pucotenlimab Combined With Lenvatinib as a Neodjuvant Therapy for Non Clear Cell Renal Cell Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, ZHOU FANGJIAN, Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-FXY-181
Record Dates: First submitted 2023-11-06; First posted 2023-11-13 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Renal Cell Carcinoma
Keywords: Pucotenlimab; Lenvatinib; Non-clear renal cell carcinoma; Neoadjuvant therapy
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — lenvatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pucotenlimab combined with Lenvatinib as neoadjuvant therapy (Experimental): Pucotenlimab combined with Lenvatinib as neoadjuvant therapy
  Interventions: Drug: Pucotenlimab Combined With Lenvatinib

INTERVENTIONS:
Drug: Pucotenlimab Combined With Lenvatinib — Patients treated by Pucotenlimab combined with Lenvatinib for 3 months before surgery

SUMMARY:
Through the neoadjuvant treatment with a combination of Pucotenlimab and Lenvatinib, it eventually enables the successful and safe implementation of partial nephrectomy in patients with localized renal cancer, who have indications for nephron-sparing surgery but face significant difficulty in kidney preservation (T1b with an endophytic component ≥75% or T2).

DETAILED DESCRIPTION:
Through the neoadjuvant treatment with a combination of Pucotenlimab and Lenvatinib, it eventually enables the successful and safe implementation of partial nephrectomy in patients with localized renal cancer, who have indications for nephron-sparing surgery but face significant difficulty in kidney preservation (T1b with an endophytic component ≥75% or T2).

ELIGIBILITY:
Inclusion Criteria:

* Voluntary signing of a written Informed Consent Form (ICF).
* Age ≥18 and <80 years at the time of enrollment, regardless of gender.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Expected survival ≥3 months.
* Preoperative biopsy confirming non-clear cell renal cancer.
* Patient's willingness to undergo nephron-sparing surgery.
* Have indications for nephron-sparing surgery but with high difficulty in kidney preservation (T1b with an endophytic component ≥75% or T2).
* At least one measurable lesion (according to mRECIST v1.1 criteria) suitable for repeated and accurate measurements.
* Good organ function, with screening laboratory results meeting the following criteria:

Hematology (no blood component or growth factor support therapy in the two weeks before treatment):

1. Absolute neutrophil count (ANC) ≥ 1.5×10^9/L (1,500/mm^3);
2. Platelet count (PLT) ≥ 100×10^9/L (100,000/mm^3);
3. Hemoglobin (HB) ≥ 90 g/L.

Hepatic function:

1. Total bilirubin (TBIL) ≤ 1.5×ULN;
2. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5×ULN; for subjects with liver metastasis, AST and ALT ≤ 5×ULN.
3. Serum albumin (ALB) ≥ 28g/L.

Coagulation function:

International normalized ratio (INR) and activated partial thromboplastin time (APTT) ≤ 1.5 × ULN.

· Willingness and ability of the subject to comply with the scheduled visits, treatment plan, laboratory tests, and other study requirements.

Exclusion Criteria:

* Renal biopsy pathology diagnosis indicates collecting duct carcinoma.
* Renal biopsy pathology diagnosis indicates chromophobe carcinoma.
* Renal biopsy pathology indicates clear cell renal cell carcinoma or predominantly clear cell renal cell carcinoma.
* Presence of lymph node metastasis.
* Tumor encases the renal artery.
* Intravascular tumor thrombus in the renal vein.
* Tumor exhibits diffuse growth without distinct boundaries from normal renal parenchyma.
* Poor general condition, unsuitable for tolerating general anesthesia surgery in anesthesia assessment.
* Severe cardiovascular or cerebrovascular disease, uncontrolled hypertension, and diabetes.
* Patients using long-term immunosuppressive agents after organ transplantation.
* Patients currently using immunosuppressive drugs.
* Patients with evident infection or fever.
* Patients with T-cell lymphoma, myeloma.
* Simultaneously having other malignant tumors, undergoing treatment for malignancies, or having a history of other malignant tumors within the past six months.
* Metastatic renal cell carcinoma.
* Received herbal or immune-modulating drugs with antitumor indications within 14 days before the first use of the investigational drug.
* Undergoing systemic therapy (excluding thoracoscopic peptide, interferon, interleukin used for controlling pleural effusion locally).
* Active or potential relapse of autoimmune diseases, except for cases not requiring systemic treatment such as stable vitiligo, alopecia, psoriasis, or eczema; hypothyroidism caused by autoimmune thyroiditis that requires stable hormone replacement therapy; Type I diabetes requiring stable insulin replacement therapy.
* Concurrent participation in another clinical study unless it is an observational, non-interventional clinical study, or the follow-up period of an interventional study.
* Known mental illness, substance abuse, alcoholism, or drug addiction history.
* Pregnant or lactating women.
* Past or current existence of any diseases, treatments, or laboratory abnormalities that might confound study results, affect the subject's full participation in the study, or participation that may not be in the subject's best interest.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Estimated)
Dates: Start 2023-11-11 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
ORR | At the end of Cycle 6 (each cycle is 14 days) of Pucotenlimab treatment
  Objective Response Rate (ORR) based on RECIST 1.1 criteria.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Other (Non U.s.), China

IPD SHARING:
Plan to Share IPD: No